CLINICAL TRIAL: NCT02656693
Title: Integrating Online Weight Management With Primary Care Support: Patient-Centered Strategies for Addressing Overweight and Obesity in Primary Care
Brief Title: Integrating Online Weight Management With Primary Care Support
Acronym: PROPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Heather J. Baer, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015P002372
Record Dates: First submitted 2016-01-04; First posted 2016-01-15 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Weight Reduction Programs; Weight Loss Programs; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Program Only (Experimental): Patients will use an online weight management program called BMIQ, with minimal additional support.
  Interventions: Behavioral: Online weight management program
- Combined Intervention (Experimental): Patients will use an online weight management program called BMIQ, but will also receive additional monitoring and support from a population health manager who works with their primary care practices.
  Interventions: Behavioral: Online weight management program; Behavioral: Population health management support
- Usual Care (No Intervention): Patients will continue receiving usual care but will also be mailed some general written information about weight management (very minimal intervention.)

INTERVENTIONS:
Behavioral: Online weight management program — Patients who are enrolled in one of the two arms using the online weight management program (BMIQ) will complete structured educational sessions, follow specific calorie goals and meal plans, participate in self-monitoring activities (i.e., regular tracking of weight, diet, and physical activity), and interact with other features of the program.
  Arms: Combined Intervention; Online Program Only
Behavioral: Population health management support — Patients will receive weight-related population health management support from their primary care practice; their online weight management program data will be monitored by the population health manager, who will conduct outreach with patients at designated points according to the protocol.
  Arms: Combined Intervention

SUMMARY:
The goal of this project is to adapt an evidence-based online weight management program and integrate it with population management support from primary care practices. Investigators then will conduct a three-arm, cluster-randomized trial to compare the effectiveness of 1) the combined intervention (online weight management program plus population management support) with 2) the stand-alone online weight management program and with 3) usual care, among overweight and obese primary care patients with type 2 diabetes or hypertension. The specific aims are:

1. a. To adapt an online weight management program and integrate it with population management support, incorporating input from patients, primary care clinicians, and other stakeholders; afterward, investigators will acquire feedback on the positive and negative aspects of the intervention.

   b. To compare the effectiveness of the combined intervention (online weight management program plus population management support) with the stand-alone online program and with usual care.

   Hypothesis 1: The combined intervention will lead to greater weight loss at 12 months compared with the stand-alone online program and with usual care.
2. To identify mediators of the combined intervention and the stand-alone online program.

   Hypothesis 2: The effects of the combined intervention and the stand-alone online program on weight loss will be mediated by patients' level of engagement, changes in self-efficacy, and changes in diet and physical activity.
3. To explore whether the effectiveness of the combined intervention and the stand-alone weight management program varies by patient characteristics.

Hypothesis 3: The interventions will be more effective among patients who are younger, white, and higher socioeconomic status, although the population management strategy may help to reduce these differences.

DETAILED DESCRIPTION:
Focus Groups and Key Informant Interviews:

Focus groups will be conducted with 5 to 7 patients at the beginning of the study to obtain their feedback about an online program and the population health management support strategy. To be eligible for the focus groups, patients must have a Brigham and Women's Hospital (BWH) primary care clinician, be between ages 20-70 years old, and have a recent BMI (in the past year) between approximately 27 and 40 kg/m2. They should also be interested in weight management and/or motivated to lose weight.

Phone interviews will be conducted at the end of the study to solicit feedback on the BMIQ program and the population health management intervention. Patients in the PROPS Study who are assigned to the online program or combined intervention arm, reach the 18-month timepoint, and complete the final study survey are eligible and will be invited to participate.

Key Informant Interviews will be conducted at the beginning and the end of the study. To be eligible, the key informants must be clinicians or other staff who provide services to patients at one of the participating BWH primary care practices. There are a total of 165 clinicians in these practices, including staff physicians, residents or fellows, and nurse practitioners or physician assistants. Approximately 7 clinicians at each timepoint will be recruited as key informants and will also be asked to complete electronic surveys during the trial.

After adapting the online weight management program and integrating it with the population management support strategy based on our focus groups and key informant interviews, investigators will conduct a three-arm cluster-randomized trial to compare the effectiveness of the combined intervention (online weight management program plus population management support) with the stand-alone online weight management program and with usual care. This will be a pragmatic clinical trial conducted in approximately 14 BWH primary care practices. To be eligible for the trial, patients must have an upcoming scheduled visit at a BWH primary care practice, BMI between 27 and 39.9 kg/m2 at enrollment, and a diagnosis of type 2 diabetes or hypertension. They also must be between ages 20 and 70 (inclusive) at enrollment, speak English or Spanish, and have access the Internet using a computer, tablet, or smart phone. Finally, patients must be motivated to lose weight. Investigators plan to recruit a total of 840 patients for the study (280 per arm). Patients who enroll in the trial will attend regular primary care visits at their practices and also will complete surveys by e-mail, regular mail, or phone.

ELIGIBILITY:
Inclusion Criteria:

1. upcoming or recent visit at primary care practice affiliated with Brigham and Women's Hospital
2. age 20-70
3. diagnosis of type 2 diabetes and/or hypertension
4. BMI >= 27 and < 40 kg/m2
5. motivated to lose weight
6. valid email address and access the Internet using a computer, tablet, or smartphone
7. English or Spanish-speaking

Exclusion Criteria:

1. on insulin for treatment of their diabetes 2. MI, stroke, or atherosclerotic cardiovascular disease (ASCVD) procedure in last 6 months 3. Unstable angina 4. Currently pregnant or planning to become pregnant during the study period 5. Currently lactating 5. Has had bariatric surgery or planning to have bariatric surgery 6. >5% weight loss in the last 6 months 7. Severe psychiatric illness or impaired mental status 8. Active or diagnosed history of and/or self-reported history of eating disorders 9. Self-reported average consumption of > 14 alcoholic drinks/week 10. Any serious medical condition that would affect weight loss or for which weight loss is contraindicated, including active cancer (excluding non-melanoma skin cancer) or currently being treated for cancer, end stage renal disease (ESRD) on dialysis, etc.

11. On comfort care measures, hospice, or in nursing home 12. Participating in a contra-indicative research study 13. Use of prescription or over-the-counter weight loss medications or an all-liquid diet program in the last 6 months or currently 14. Any other medical contraindication for weight loss or physical activity, or any other reason that the PCP or their delegate (e.g., LPN or RN) did not deem the patient appropriate for the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Baer, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baer HJ, Rozenblum R, De La Cruz BA, Orav EJ, Wien M, Nolido NV, Metzler K, McManus KD, Halperin F, Aronne LJ, Minero G, Block JP, Bates DW. Effect of an Online Weight Management Program Integrated With Population Health Management on Weight Change: A Randomized Clinical Trial. JAMA. 2020 Nov 3;324(17):1737-1746. doi: 10.1001/jama.2020.18977. PMID 33141209
- [Derived] Baer HJ, De La Cruz BA, Rozenblum R, Nolido NV, Orav EJ, Metzler K, Block JP, Halperin F, McManus KD, Aronne LJ, Minero G, Bates DW. Integrating an online weight management program with population health management in primary care: Design, methods, and baseline data from the PROPS randomized controlled trial (Partnerships for Reducing Overweight and Obesity with Patient-centered Strategies). Contemp Clin Trials. 2020 Aug;95:106026. doi: 10.1016/j.cct.2020.106026. Epub 2020 May 16. PMID 32428586
- [Derived] Rozenblum R, De La Cruz BA, Nolido NV, Adighibe I, Secinaro K, McManus KD, Halperin F, Block JP, Bates DW, Baer HJ. Primary Care Patients' and Providers' Perspectives about an Online Weight Management Program: a Qualitative Study. J Gen Intern Med. 2019 Aug;34(8):1503-1521. doi: 10.1007/s11606-019-05022-6. Epub 2019 May 31. PMID 31152361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Started | 326 | 216 | 298
Completed | 325 | 214 | 295
Not Completed | 1 | 2 | 3
Not completed — Pregnancy | 1 | 1 | 1
Not completed — Bariatric surgery | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Online Program Only | Combined Intervention | Total
Number analyzed (Participants) | 326 | 216 | 298 | 840
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (8.6) | 59.1 (8.8) | 60.1 (8.3) | 59.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 128 | 159 | 504
  Male | 109 | 88 | 139 | 336
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because missing data has been excluded from this table.
  Participants
    number analyzed (Participants) | 326 | 215 | 295 | 836
    White, non-Hispanic | 249 | 169 | 227 | 645
    Black, non-Hispanic | 39 | 23 | 31 | 93
    Hispanic | 24 | 12 | 20 | 56
    Other/multiple categories | 14 | 11 | 17 | 42
Weight [Mean (Standard Deviation); unit: kgs] | 91.8 (14.4) | 91.6 (14.4) | 92.9 (13.8) | 92.1 (14.3)
Height [Mean (Standard Deviation); unit: centimeters] | 167.4 (9.4) | 168.7 (9.9) | 169.2 (9.9) | 168.4 (9.9)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (3.3) | 32.2 (3.2) | 32.4 (3.4) | 32.5 (3.3)
Medical conditions [Count of Participants; unit: Participants]
  Hypertension | 312 | 211 | 287 | 810
  Type 2 diabetes | 73 | 49 | 83 | 205
  Hypercholesterolemia | 67 | 60 | 56 | 183
  Obstructive sleep apnea | 53 | 36 | 56 | 145
  Coronary heart disease/ atherosclerosis | 2 | 1 | 4 | 7
  Non-alcoholic fatty liver disease | 1 | 1 | 3 | 5
Highest level of education [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because missing data has been excluded from this table.
  Participants
    number analyzed (Participants) | 288 | 192 | 258 | 738
    High school graduate or less | 23 | 16 | 14 | 53
    Some college | 91 | 45 | 50 | 186
    College graduate | 102 | 66 | 83 | 251
    Master's, doctorate, or professional degree | 72 | 65 | 111 | 248
Employment status [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because missing data has been excluded from this table.
  Participants
    number analyzed (Participants) | 314 | 213 | 288 | 815
    Employed (full-time or part-time) | 206 | 139 | 169 | 514
    Retired | 63 | 33 | 65 | 161
    Other | 45 | 41 | 54 | 140
Health insurance [Count of Participants; unit: Participants]
  Private | 217 | 141 | 207 | 565
  Medicare | 72 | 50 | 68 | 190
  Medicaid/VA | 37 | 25 | 23 | 85
Any previous weight loss attempts [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because missing data has been excluded from this table.
  Participants
    number analyzed (Participants) | 291 | 188 | 266 | 745
    (all) | 269 | 182 | 236 | 687
Motivation to lose weight [Mean (Standard Deviation); unit: scores on a scale] — During the screening process, participants were asked about their motivation to lose weight in the next 6 months, using a 10-point Likert scale where 1= not at all motivated and 10= completely or extremely motivated. This simple measure has been used in previous studies and is associated with behavior change. Only patients who report their level of motivation to be 7 or higher were eligible to participate in the study.
  scores on a scale | 8.8 (1.1) | 8.9 (1.1) | 8.9 (1.1) | 8.9 (1.1)
Internet use [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because missing data has been excluded from this table.
  Participants
    number analyzed (Participants) | 287 | 191 | 260 | 738
    </= Once per week | 6 | 2 | 4 | 12
    Several times per week | 14 | 13 | 8 | 35
    Once per day | 23 | 9 | 14 | 46
    >/= Several times per day | 244 | 167 | 234 | 645
Primary language [Count of Participants; unit: Participants]
  English | 315 | 212 | 288 | 815
  Spanish | 11 | 4 | 10 | 25
Use of GLP-1 receptor agonist of SGLT2 inhibitors [Count of Participants; unit: Participants] | 1 | 1 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight at 12 Months
Description: change in body weight from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
kilograms | -1.2 [-2.1 to -0.3] | -1.9 [-2.6 to -1.1] | -3.1 [-3.7 to -2.5]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.00017, Mixed Models Analysis

2. Secondary Outcome: Change in Body Weight at 6 Months
Description: change in body weight from enrollment to 6 months
Time Frame: 6 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
kilograms | -1.0 [-1.9 to -0.1] | -2.1 [-2.8 to -1.5] | -2.9 [-3.5 to -2.3]

3. Secondary Outcome: Change in Body Weight at 18 Months
Description: change in body weight from enrollment to 18 months
Time Frame: 18 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
kilograms | -1.9 [-2.8 to -1.0] | -1.1 [-2.0 to -0.3] | -2.8 [-3.5 to -2.0]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Percent Weight Change at 6 Months
Description: Percent weight change from enrollment to 6 months
Time Frame: 6 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of weight change
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of weight change | -1.0 [-1.9 to 0.03] | -2.0 [-3.1 to -0.9] | -2.8 [-3.8 to -1.8]

5. Secondary Outcome: Percent Weight Change at 12-Months
Description: Percent weight change from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of weight change
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of weight change | -1.4 [-2.3 to -0.6] | -1.9 [-2.8 to -1.0] | -3.0 [-3.8 to -2.1]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: Percent Weight Change at 18-Months
Description: Percent weight change from enrollment to 18 months
Time Frame: 18 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of weight change
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of weight change | -1.9 [-2.9 to -0.9] | -0.9 [-2.0 to 0.2] | -2.6 [-3.6 to -1.5]
Statistical Analysis 1: Comparison: Usual Care vs Combined Intervention; Test type: Superiority; p = 0.01, Mixed Models Analysis

7. Secondary Outcome: Percent of Patients With at Least 5% Weight Loss at 6 Months
Description: Percent of Patients With at Least 5% Weight Loss from enrollment to 6 months
Time Frame: 6-months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of patients | 13.4 [7.8 to 19.0] | 22.1 [14.2 to 30.0] | 29.5 [21.4 to 37.5]

8. Secondary Outcome: Percent of Patients With at Least 5% Weight Loss at 12-months
Description: Percent of Patients with at least 5% weight loss from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of patients | 14.9 [10.2 to 19.6] | 20.8 [14.5 to 27.2] | 32.3 [25.8 to 38.8]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis

9. Secondary Outcome: Percent of Patients With at Least 5% Weight Loss at 18 Months
Description: Percent of Patients With at least 5% weight loss from enrollment to 18 months
Time Frame: 18-months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: percentage of patients
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of patients | 20.9 [14.3 to 27.6] | 19.9 [12.5 to 27.3] | 31.3 [23.0 to 39.6]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.20, Mixed Models Analysis

10. Secondary Outcome: Changes in Self-efficacy Around Weight Loss at 12 Months
Description: Changes in self-efficacy around weight loss at 12 months Self-efficacy will be assessed by asking patients to rate their confidence in their ability to lose weight on a scale from 1 ("not at all confident") to 10 ("very confident"). A rank of 1-7 reflects low self-efficacy, while 8-10 reflects high self-efficacy based on Bandura's theory of self-efficacy.
Time Frame: 12 months after initial primary care visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
score on a scale | -0.7 [-1.1 to -0.3] | -0.4 [-0.9 to 0.07] | 0.5 [0.06 to 0.9]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.0001, Mixed Models Analysis

11. Secondary Outcome: Changes in Systolic Blood Pressure
Description: changes in systolic blood pressure (BP) from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mmHg | -0.9 [-2.8 to 1.0] | -3.0 [-5.4 to -0.6] | -0.2 [-2.3 to 1.9]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.19, Mixed Models Analysis

12. Secondary Outcome: Changes in Diastolic Blood Pressure
Description: changes in diastolic blood pressure (BP) from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mmHg | -1.0 [-2.2 to 0.3] | -2.2 [-3.8 to -0.7] | -1.1 [-2.4 to 0.2]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.35, Mixed Models Analysis

13. Secondary Outcome: Changes in Total Cholesterol
Description: changes in total cholesterol from Enrollment to 12 Months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mg/dL | -7.5 [-13.2 to -1.8] | -6.3 [-13.4 to 0.9] | -6.8 [-12.4 to -1.1]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.20, Mixed Models Analysis

14. Secondary Outcome: Changes in HDL Cholesterol
Description: changes in HDL cholesterol from Enrollment to 12 Months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mg/dL | -0.4 [-2.2 to 1.3] | 0.6 [-1.8 to 3.1] | 0.7 [-1.3 to 2.7]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.33, Mixed Models Analysis

15. Secondary Outcome: Changes in LDL Cholesterol
Description: changes in LDL cholesterol from Enrollment to 12 Months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mg/dL | -5.4 [-10.1 to -0.7] | -3.7 [-9.2 to 1.8] | -5.8 [-10.3 to -1.2]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.43, Mixed Models Analysis

16. Secondary Outcome: Changes in Triglycerides
Description: changes in triglycerides from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
mg/dL | -12.4 [-24.9 to 0.06] | -8.0 [-24.2 to 8.1] | -10.2 [-23.5 to 3.1]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.40, Mixed Models Analysis

17. Secondary Outcome: Changes in HbA1c Levels
Description: changes in Hemoglobin (HbA1c) levels from enrollment to 12 months
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: % of HbA1c
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
% of HbA1c | -0.02 [-0.1 to 0.1] | 0.02 [-0.1 to 0.2] | -0.02 [-0.2 to 0.1]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.16, Mixed Models Analysis

18. Secondary Outcome: Changes in Weight-related Quality of Life Assessed by the Impact of Weight on Quality of Life (IWQOL)-Lite Questionnaire
Description: Weight-related quality of life will be assessed using the Impact of Weight of Quality of Life (IWQOL)-Lite questionnare. The IWQOL-Lite is a brief, 31-item self-report measure that consists of scores on five scales (physical function, self-esteem, sexual life, public distress, and work) and a total score (sum of scale scores). Participants are asked to rate items with respect to the past week, with responses from "never true" to "always true". Total scores range from 0 (worst possible quality of life) to 100 (best possible quality of life).
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
score on a scale | 5.4 [4.0 to 6.8] | 4.8 [3.0 to 6.7] | 5.8 [4.2 to 7.4]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.61, Mixed Models Analysis

19. Secondary Outcome: Changes in Percentage of Patients Reporting Excellent/Very Good Health Status Assessed by Using a 5-point Scale Questionnaire From the 36-Item Short Form Health Survey(SF-36)
Description: Health status will be assessed using 5-point scale response to a single question from the SF-36, "In general, would you say that your health is...(1=Excellent, 2=Very Good, 3=Good, 4=Fair, 5=Poor"). A higher score indicates a worse outcome (5= poor health status).
Time Frame: 12 months after the initial primary care visit
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
percentage of patients | 14.5 [6.0 to 23.1] | 16.1 [4.8 to 27.4] | 21.4 [12.7 to 30.0]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.61, Mixed Models Analysis

20. Secondary Outcome: Changes in Self-reported Physical Activity
Description: changes in self-reported physical activity minutes per week
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: minutes/week
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
minutes/week | 5.7 [-1.3 to 12.7] | 2.6 [-6.8 to 12.0] | 3.5 [-3.7 to 10.7]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.46, Mixed Models Analysis

21. Secondary Outcome: Changes in Diet, Specifically Fruits/Vegetables, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically fruits/vegetables as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | 0.4 [0.2 to 0.6] | 0.3 [0.04 to 0.7] | 0.4 [0.2 to 0.7]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.68, Mixed Models Analysis

22. Secondary Outcome: Changes in Diet, Specifically Whole Grains, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically whole grains as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | 0.02 [-0.05 to 0.1] | 0.03 [-0.07 to 0.1] | 0.1 [0.01 to 0.2]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.54, Mixed Models Analysis

23. Secondary Outcome: Changes in Diet, Specifically Sugar-sweetened Beverages, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically sugar-sweetened beverages as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | 0.01 [-0.05 to 0.08] | -0.1 [-0.2 to 0.01] | -0.1 [-0.1 to 0.01]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.09, Mixed Models Analysis

24. Secondary Outcome: Changes in Diet, Specifically Baked Products, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically baked products as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | -0.1 [-0.1 to -0.02] | -0.1 [-0.1 to 0.02] | -0.1 [-0.1 to -0.003]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.42, Mixed Models Analysis

25. Secondary Outcome: Changes in Diet, Specifically Processed Meats, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically processed meats as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | -0.02 [-0.1 to 0.02] | -0.1 [-0.1 to -0.01] | -0.1 [-0.1 to -0.01]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.23, Mixed Models Analysis

26. Secondary Outcome: Changes in Diet, Specifically Fried Foods, as Measured by the PrimeScreen Questionnaire
Description: changes in diet, specifically fried foods as measured by the PrimeScreen questionnaire, a brief dietary screening tool.
Time Frame: 12 months after the initial primary care visit
Measure: Mean (95% Confidence Interval); unit: servings/day
Arm/Group | Usual Care | Online Program Only | Combined Intervention
Number analyzed (Participants) | 326 | 216 | 298
servings/day | -0.03 [-0.1 to 0.01] | -0.02 [-0.1 to 0.03] | -0.1 [-0.1 to -0.02]
Statistical Analysis 1: Comparison: Usual Care vs Online Program Only vs Combined Intervention; Test type: Superiority; p = 0.20, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of enrollment to 18 months (+/- 90 days) after enrollment in the study.
Description: Staff received "research notifications" via the electronic health record whenever enrolled patients were admitted to and/or seen in the Emergency Dept of any Partners-affiliated hospital. Participants were also encouraged to self-report any serious medical conditions. Cases were regularly reviewed by research staff and escalated to the Principal Investigator, co-investigators, and patients' PCPs, as needed. Adverse events were reported/documented per Partners IRB guidelines.
Arm/Group | Usual Care | Online Program Only | Combined Intervention
All-Cause Mortality (participants affected / at risk) | 0/326 | 0/216 | 1/298
Serious Adverse Events (participants affected / at risk) | 12/326 | 11/216 | 18/298
Other Adverse Events (participants affected / at risk) | 0/326 | 0/216 | 0/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=326) | Online Program Only (N=216) | Combined Intervention (N=298)
Angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary arteriogram (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass grafting (CABG) (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart attack (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 3 (3)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Brain surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis of lumbar region (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Transient ischemic attack (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02656693/Prot_SAP_000.pdf